CLINICAL TRIAL: NCT05660525
Title: Leveraging Community Pharmacists to Optimize Smoking Cessation Services for Rural Smokers in Appalachia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Melissa Little, PhD, MPH, Associate Professor, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HSR220197
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Smoking Cessation; Smoking, Cigarette; Smoking Reduction; Smoking; Smoking, Tobacco; Quitting Smoking
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking; Smoking Reduction; Smoking; Tobacco Smoking | interventions — Tobacco Use Cessation Devices; Medication Therapy Management

STUDY DESIGN:
Intervention Model Description: 2x2x2x2x2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (32):
- QuitAid, 4 weeks, Patch + Lozenge (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist and 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and the nicotine lozenge.
  Interventions: Drug: 4 weeks of Nicotine lozenge; Behavioral: QuitAid; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- QuitAid, 8 weeks, Patch + Lozenge (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist and 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and the nicotine lozenge.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: QuitAid; Drug: 8 Weeks Nicotine Lozenge
- QuitAid, 4 weeks, Patch + Lozenge, QuitLine (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and the nicotine lozenge, and a Quitline intervention
  Interventions: Drug: 4 weeks of Nicotine lozenge; Behavioral: QuitAid; Behavioral: Tobacco Quitline; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- QuitAid, 8 weeks, Patch + Lozenge, QuitLine (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and the nicotine lozenge, and a Quitline intervention
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: QuitAid; Behavioral: Tobacco Quitline; Drug: 8 Weeks Nicotine Lozenge
- QuitAid, 4 weeks, Patch (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist and 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch.
  Interventions: Behavioral: QuitAid; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- QuitAid, 8 weeks, Patch (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist and 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: QuitAid
- QuitAid, 8 weeks, Patch, QuitLine (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch, and a Quitline intervention
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: QuitAid; Behavioral: Tobacco Quitline
- QuitAid, 4 weeks, Patch, QuitLine (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch, and a Quitline intervention
  Interventions: Behavioral: QuitAid; Behavioral: Tobacco Quitline; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- QuitAid, 4 weeks, Patch, SmokeFree Txt (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch, and a texting intervention to help quit smoking.
  Interventions: Behavioral: QuitAid; Behavioral: Smokefree TXT; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- QuitAid, 8 weeks, Patch, SmokeFree Txt (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch, and a texting intervention to help quit smoking.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: QuitAid; Behavioral: Smokefree TXT
- QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge, and a texting intervention to help quit smoking.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: QuitAid; Behavioral: Smokefree TXT; Drug: 8 Weeks Nicotine Lozenge
- QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge, and a texting intervention to help quit smoking.
  Interventions: Drug: 4 weeks of Nicotine lozenge; Behavioral: QuitAid; Behavioral: Smokefree TXT; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge, a texting intervention to help quit smoking, and a Quitline Intervention.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: QuitAid; Behavioral: Smokefree TXT; Behavioral: Tobacco Quitline; Drug: 8 Weeks Nicotine Lozenge
- QuitAid, 8 weeks, Patch, SmokeFree Txt, QuitLine (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch, a texting intervention to help quit smoking, and a Quitline Intervention.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: QuitAid; Behavioral: Smokefree TXT; Behavioral: Tobacco Quitline
- QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge, a texting intervention to help quit smoking, and a Quitline Intervention.
  Interventions: Drug: 4 weeks of Nicotine lozenge; Behavioral: QuitAid; Behavioral: Smokefree TXT; Behavioral: Tobacco Quitline; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- QuitAid, 4 weeks, Patch, SmokeFree Txt, QuitLine (Experimental): Smoking participants receive QuitAid, a medication therapy management delivered by their pharmacist, 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch, a texting intervention to help quit smoking, and a Quitline Intervention.
  Interventions: Behavioral: QuitAid; Behavioral: Smokefree TXT; Behavioral: Tobacco Quitline; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine (Experimental): Smoking participants receive 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge, a texting intervention to help quit smoking, and a Quitline Intervention.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: Smokefree TXT; Behavioral: Tobacco Quitline; Drug: 8 Weeks Nicotine Lozenge
- 8 weeks, Patch, SmokeFree Txt, QuitLine (Experimental): Smoking participants receive 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch, a texting intervention to help quit smoking, and a Quitline Intervention.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: Smokefree TXT; Behavioral: Tobacco Quitline
- 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine (Experimental): Smoking participants receive 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge, a texting intervention to help quit smoking, and a Quitline Intervention.
  Interventions: Drug: 4 weeks of Nicotine lozenge; Behavioral: Smokefree TXT; Behavioral: Tobacco Quitline; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- 4 weeks, Patch, SmokeFree Txt, QuitLine (Experimental): Smoking participants receive 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch, a texting intervention to help quit smoking, and a Quitline Intervention.
  Interventions: Behavioral: Smokefree TXT; Behavioral: Tobacco Quitline; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- 8 weeks, Patch + Lozenge, QuitLine (Experimental): Smoking participants receive 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge, and a Quitline Intervention.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: Tobacco Quitline; Drug: 8 Weeks Nicotine Lozenge
- 8 weeks, Patch, QuitLine (Experimental): Smoking participants receive 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch, and a Quitline Intervention.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: Tobacco Quitline
- 4 weeks, Patch + Lozenge, QuitLine (Experimental): Smoking participants receive 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge, and a Quitline Intervention.
  Interventions: Drug: 4 weeks of Nicotine lozenge; Behavioral: Tobacco Quitline; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- 4 weeks, Patch, QuitLine (Experimental): Smoking participants receive 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch, and a Quitline Intervention.
  Interventions: Behavioral: Tobacco Quitline; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- 8 weeks, Patch + Lozenge, SmokeFree Txt (Experimental): Smoking participants receive 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge and a texting intervention to help quit smoking.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: Smokefree TXT; Drug: 8 Weeks Nicotine Lozenge
- 8 weeks, Patch, SmokeFree Txt (Experimental): Smoking participants receive 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and a texting intervention to help quit smoking.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Behavioral: Smokefree TXT
- 4 weeks, Patch + Lozenge, SmokeFree Txt (Experimental): Smoking participants receive 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge and a texting intervention to help quit smoking.
  Interventions: Drug: 4 weeks of Nicotine lozenge; Behavioral: Smokefree TXT; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- 4 weeks, Patch, SmokeFree Txt (Experimental): Smoking participants receive 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and a texting intervention to help quit smoking.
  Interventions: Behavioral: Smokefree TXT; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- 8 weeks, Patch + Lozenge (Experimental): Smoking participants receive 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch; Drug: 8 Weeks Nicotine Lozenge
- 8 weeks, Patch (Experimental): Smoking participants receive 8 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch.
  Interventions: Drug: 8 weeks of Nicotine Replacement Therapy Patch
- 4 weeks, Patch + Lozenge (Experimental): Smoking participants receive 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch and lozenge.
  Interventions: Drug: 4 weeks of Nicotine lozenge; Drug: 4 weeks of Nicotine Replacement Therapy Patch
- 4 weeks, Patch (Experimental): Smoking participants receive 4 weeks Nicotine Replacement Therapy (NRT) in the form of the nicotine patch.
  Interventions: Drug: 4 weeks of Nicotine Replacement Therapy Patch

INTERVENTIONS:
Drug: 4 weeks of Nicotine lozenge — All participants will receive at least 4 weeks of the NRT Patch. Some will be randomized to receive 4 weeks of lozenge in addition to the NRT Patch. NRT temporarily replaces nicotine from tobacco to reduce motivation to consume tobacco and nicotine withdrawal symptoms.
  Other Names: Sunmark Nicotine Polacrilex Lozenge; Habitrol Nicotine Lozenge; Nicotinell Nicotine Lozenge; Nicorette Lozenge
  Arms: 4 weeks, Patch + Lozenge; 4 weeks, Patch + Lozenge, QuitLine; 4 weeks, Patch + Lozenge, SmokeFree Txt; 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; QuitAid, 4 weeks, Patch + Lozenge; QuitAid, 4 weeks, Patch + Lozenge, QuitLine; QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt; QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine
Drug: 8 weeks of Nicotine Replacement Therapy Patch — All participants will receive at least 4 weeks of the NRT Patch. Some will also be randomized to receive an additional 4 weeks of the NRT Patch
  Other Names: Habitrol Transdermal Product; Pixotine Transdermal Product; Lucy Transdermal Product; Nicoderm C-Q Transdermal Product; Nicotrol Transdermal Product
  Arms: 8 weeks, Patch; 8 weeks, Patch + Lozenge; 8 weeks, Patch + Lozenge, QuitLine; 8 weeks, Patch + Lozenge, SmokeFree Txt; 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; 8 weeks, Patch, QuitLine; 8 weeks, Patch, SmokeFree Txt; 8 weeks, Patch, SmokeFree Txt, QuitLine; QuitAid, 8 weeks, Patch; QuitAid, 8 weeks, Patch + Lozenge; QuitAid, 8 weeks, Patch + Lozenge, QuitLine; QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt; QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; QuitAid, 8 weeks, Patch, QuitLine; QuitAid, 8 weeks, Patch, SmokeFree Txt; QuitAid, 8 weeks, Patch, SmokeFree Txt, QuitLine
Behavioral: QuitAid — All participants will receive at least 4 weeks of the NRT Patch. Some participants will also be randomized to receive the QuitAid intervention, based on a medication adherence intervention, addresses perceptions (e.g., motivation, self-efficacy, beliefs) and practicalities of using NRT (e.g., monitoring NRT use, establishing a reminder system). QuitAid includes 1 in-person session and 5 follow-up telephonic sessions with the participant's local pharmacist/technician.
  Other Names: Medication Therapy Management (MTM)
  Arms: QuitAid, 4 weeks, Patch; QuitAid, 4 weeks, Patch + Lozenge; QuitAid, 4 weeks, Patch + Lozenge, QuitLine; QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt; QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; QuitAid, 4 weeks, Patch, QuitLine; QuitAid, 4 weeks, Patch, SmokeFree Txt; QuitAid, 4 weeks, Patch, SmokeFree Txt, QuitLine; QuitAid, 8 weeks, Patch; QuitAid, 8 weeks, Patch + Lozenge; QuitAid, 8 weeks, Patch + Lozenge, QuitLine; QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt; QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; QuitAid, 8 weeks, Patch, QuitLine; QuitAid, 8 weeks, Patch, SmokeFree Txt; QuitAid, 8 weeks, Patch, SmokeFree Txt, QuitLine
Behavioral: Smokefree TXT — All participants will receive at least 4 weeks of the NRT Patch. Some participants will also be randomized to receive the SmokefreeTXT is a text-messaging program offered through the National Cancer Institute's Smokefree.gov initiative, which sends pre-programmed messages timed around a quit date. Participants will receive 3-5 messages a day for 7 weeks. The first week of messages focus on preparation and the remaining 6 weeks of messages focus on post-cessation strategies (e.g., relapse prevention), all timed relative to the quit date set at enrollment.
  Arms: 4 weeks, Patch + Lozenge, SmokeFree Txt; 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; 4 weeks, Patch, SmokeFree Txt; 4 weeks, Patch, SmokeFree Txt, QuitLine; 8 weeks, Patch + Lozenge, SmokeFree Txt; 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; 8 weeks, Patch, SmokeFree Txt; 8 weeks, Patch, SmokeFree Txt, QuitLine; QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt; QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; QuitAid, 4 weeks, Patch, SmokeFree Txt; QuitAid, 4 weeks, Patch, SmokeFree Txt, QuitLine; QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt; QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; QuitAid, 8 weeks, Patch, SmokeFree Txt; QuitAid, 8 weeks, Patch, SmokeFree Txt, QuitLine
Behavioral: Tobacco Quitline — All participants will receive at least 4 weeks of the NRT Patch. Some participants will also be randomized to receive a 4-session proactive tobacco quitline, with each session lasting 20-30 minutes and occurring on days 7, 14, 21 and 28.The quitline intervention incorporates 3 phases: (1) preparing to quit, (2) quitting process, and (3) relapse prevention.
  Arms: 4 weeks, Patch + Lozenge, QuitLine; 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; 4 weeks, Patch, QuitLine; 4 weeks, Patch, SmokeFree Txt, QuitLine; 8 weeks, Patch + Lozenge, QuitLine; 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; 8 weeks, Patch, QuitLine; 8 weeks, Patch, SmokeFree Txt, QuitLine; QuitAid, 4 weeks, Patch + Lozenge, QuitLine; QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; QuitAid, 4 weeks, Patch, QuitLine; QuitAid, 4 weeks, Patch, SmokeFree Txt, QuitLine; QuitAid, 8 weeks, Patch + Lozenge, QuitLine; QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; QuitAid, 8 weeks, Patch, QuitLine; QuitAid, 8 weeks, Patch, SmokeFree Txt, QuitLine
Drug: 4 weeks of Nicotine Replacement Therapy Patch — All participants will receive at least 4 weeks of the NRT Patch.
  Other Names: Nicotrol Transdermal Product; Nicoderm C-Q Transdermal Product; Lucy Transdermal Product; Pixotine Transdermal Product; Habitrol Transdermal Product
  Arms: 4 weeks, Patch; 4 weeks, Patch + Lozenge; 4 weeks, Patch + Lozenge, QuitLine; 4 weeks, Patch + Lozenge, SmokeFree Txt; 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; 4 weeks, Patch, QuitLine; 4 weeks, Patch, SmokeFree Txt; 4 weeks, Patch, SmokeFree Txt, QuitLine; QuitAid, 4 weeks, Patch; QuitAid, 4 weeks, Patch + Lozenge; QuitAid, 4 weeks, Patch + Lozenge, QuitLine; QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt; QuitAid, 4 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; QuitAid, 4 weeks, Patch, QuitLine; QuitAid, 4 weeks, Patch, SmokeFree Txt; QuitAid, 4 weeks, Patch, SmokeFree Txt, QuitLine
Drug: 8 Weeks Nicotine Lozenge — All participants will receive at least 4 weeks of the NRT Patch. Some will be randomized to receive 8 weeks of lozenge in addition to the NRT Patch. NRT temporarily replaces nicotine from tobacco to reduce motivation to consume tobacco and nicotine withdrawal symptoms.
  Other Names: Sunmark Nicotine Polacrilex Lozenge; Habitrol Nicotine Lozenge; Nicotinell Nicotine Lozenge; Nicorette Lozenge
  Arms: 8 weeks, Patch + Lozenge; 8 weeks, Patch + Lozenge, QuitLine; 8 weeks, Patch + Lozenge, SmokeFree Txt; 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine; QuitAid, 8 weeks, Patch + Lozenge; QuitAid, 8 weeks, Patch + Lozenge, QuitLine; QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt; QuitAid, 8 weeks, Patch + Lozenge, SmokeFree Txt, QuitLine

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and implementation of a pharmacist-delivered MTM (medication therapy management) approach, called QuitAid, to quitting cigarette smoking in rural Appalachia.

The main questions it aims to answer are:

* Is QuitAid, alone or combined with other quitting tobacco treatments, effective?
* What makes QuitAid easy or hard to carry out? Is it cost effective? Is it easy to maintain?

Treatment:

All participants will be given at least 4 weeks of the nicotine patch.

Some participants will be randomized (like the flip of a coin) to receive additional treatments (listed below).

These groups will be compared to each other to see which combination works best to help them quit smoking.

* Smokefree TXT - a texting program that helps people quit smoking
* Tobacco quitline - 4 phone sessions to help people quit smoking
* 8 weeks of NRT (nicotine replacement therapy in the form of nicotine patches or nicotine patches and lozenge) medication instead of 4 weeks
* QuitAid - An MTM program given by the patient's pharmacist. This is a quitting smoking coaching program
* Nicotine patch AND nicotine lozenge instead of just nicotine patches

DETAILED DESCRIPTION:
The proposed study uses a mixed-method design to evaluate the effectiveness and implementation of a pharmacist-delivered MTM (Medication Therapy Management) approach, called QuitAid, to smoking cessation in rural Appalachia. Aim 1 of this project will evaluate the effectiveness of QuitAid and standard, evidence-based tobacco treatments on cessation within an MTM pharmacist-delivered approach. Aim 2 will assess implementation, including relative cost of QuitAid, as well as standard, evidence-based tobacco treatments through an ask-advise-connect model, in community pharmacies, and will examine facilitators and barriers to reach, adoption, and maintenance of QuitAid as well as standard, evidence-based tobacco treatments through an ask-advise-connect method in community pharmacies.

Smokers (n=768) recruited through 14 community pharmacies in rural Appalachia will be randomized in a 2x2x2x2x2 full factorial experiment to the following five treatments: (1) QuitAid Intervention (Yes vs. No), (2) tobacco quitline (Yes vs. No), (3) SmokefreeTXT through the National Cancer Institute's (NCI) Smokefree.gov initiative (Yes vs. No), (4) Combination NRT Lozenge + NRT Patch (vs. NRT patch alone), and/or (5) 8 weeks of NRT (vs. standard 4 weeks). Following the experimental trial, we will use an implementation science approach to assess implementation, including relative cost, as well as facilitators and barriers of reach, adoption, and maintenance of QuitAid and standard, evidence-based tobacco treatments through an ask-advise-connect method in community pharmacies (Aim 2).

ELIGIBILITY:
Study participants will be rural cigarette smokers from Virginia, Tennessee, Kentucky and North Carolina who visit one of the participating study pharmacies. Pharmacies will be located in rural geographic areas of the Central and South Central subregions of Appalachia that include Virginia, Tennessee, Kentucky and North Carolina, as defined by the USDA Rural-Urban Continuum Codes (RUCC) 4-9, Rural-Urban Commuting Area (RUCA) codes 4-10, or Frontier and Remote (FAR) areas level 4. No exclusionary criteria are based on race, gender, or age.

Inclusion Criteria include:

* must be 18 years of age and older
* must be able to read, speak, and understand English
* must report smoking at least 5 cigarettes per day for the past 6 months (regardless of non-cigarette tobacco product use)
* must be willing to set a quit date within the next 30 days
* must own a cell phone
* must be willing and able to use NRT in the form of patch or lozenge
* Not be pregnant or planning to be pregnant in the next 6 months.

Exclusion Criteria include:

* are pregnant women (self-reported), breastfeeding, planning to become pregnant during the next 6 months
* have a medical contraindication to NRT (e.g., past 30 days, heart attack or stroke; past 6 months, serious or worsening angina, very rapid or irregular heartbeat requiring medication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 768 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Tobacco Abstinence | 6 months
  The primary outcome is biochemically verified point prevalence (verified through a CO test via Smokerlyzer at endpoint of participation in trial) abstinence defined as no smoking (even a puff) within the past 7 days.

SECONDARY OUTCOMES:
Self-Reported Tobacco Abstinence | 1, 2, and 3 months
  Self-reported point prevalence abstinence defined as no smoking (even a puff) within the past 7 days
Adherence to assigned treatment components | 1, 2, and 3 months
  Assess adherence to assigned treatment regimen as the percentage of sessions completed if the participant was assigned to QuitAid and/or the quitline treatments, the frequency of opt-out from SmokefreeTXT (e.g., texting "STOP"), and the percent of NRT used. Adherence to NRT (both patch and/or lozenge) will be collected from participants at the 1-, 2-, and 3-month follow-ups.
Quit Attempts | 1, 2, and 3 months
  Assess the number of times that participants have made a quit attempt since the previous contact at the 1-, 2-, 3- and 6-month follow-ups. A "quit attempt" will be defined as cigarette abstinence for ≥ 24 hours not due to involuntary or forced cessation (i.e., hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Little, PhD, MPH, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share data at the individual level

REFERENCES:
- [Derived] Fahey MC, Krukowski RA, Anderson RT, Cohn WF, Porter KJ, Reid T, Wiseman KP, You W, Wood CH, Rucker TW, Little MA. Reaching adults who smoke cigarettes in rural Appalachia: Rationale, design & analysis plan for a mixed-methods study disseminating pharmacy-delivered cessation treatment. Contemp Clin Trials. 2023 Nov;134:107335. doi: 10.1016/j.cct.2023.107335. Epub 2023 Sep 18. PMID 37730197